CLINICAL TRIAL: NCT01545427
Title: A Proof of Concept Trial of Gleevec (Imatinib) in Active Diffuse Scleroderma
Brief Title: Proof of Concept Trial of Gleevec (Imatinib) in Active Diffuse Scleroderma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Frequent adverse events occurred early in treatment with poor tolerability.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Janet Pope, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-07-214; #031-06 (Other Grant/Funding Number: Lawson Health Research Institute Internal Research Fund)
Record Dates: First submitted 2012-03-01; First posted 2012-03-06 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Scleroderma
Keywords: Scleroderma; Randomized controled trial; Pilot study; Gleevec (imatinib); Biomarkers
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Imatinib Mesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gleevec (Experimental): Gleevec 200 mg bid for 6 months.
  Interventions: Drug: Imatinib mesylate
- Placebo (Placebo Comparator): Placebo coated to appear identical to Gleevec.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Imatinib mesylate — 200 mg bid for 6 months
  Other Names: Gleevec
  Arms: Gleevec
Other: Placebo — Placebo coated to match appearance of Gleevec identically.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effectiveness and safety of the drug Gleevec (imatinib) as a new treatment for patients with active diffuse scleroderma. This drug has not been used previously to treat scleroderma, but it has been found to advance the treatment and life span of patients with a type of leukemia called chronic myeloid leukemia or CML. Gleevec acts on chemical signals in the cells that may decrease fibrosis (the hardening of the skin that occurs in scleroderma). It works by interfering in the process that activates many molecules that cause fibrosis, including TGFbeta (which may be a key part of disease activity in scleroderma).

This study proposes to treat patients that have significant diffuse scleroderma with Gleevec for 6 months and investigate several measures of scleroderma disease activity before, during and at the end of treatment (0, 3 months and 6 months). This is a randomized, double blind, placebo-controlled trial: 20 patients will be divided into two groups in a 4:1 ratio, with 16 patients taking 400mg of Gleevec per day and 4 taking a placebo. The differences between the groups that will be measured include safety, Modified Rodnan skin score (mRSS), Health Assessment Questionnaire (HAQ), global assessments (100mm VAS) and changes in biomarkers in blood and skin biopsies.

DETAILED DESCRIPTION:
Purpose:

Scleroderma is a connective tissue disease that is prototypical for fibrosis with autoantibodies and vascular abnormalities including vasomotor instability (Raynaud's) at one end and blood vessel obliteration at the other (1,2). Scleroderma occurs in > 2/10,000 (with thousands of Canadians affected) and has no proven therapy to modify the disease overall (3). The purpose of this study is to investigate the potential of Gleevec to be used as a novel therapy in the treatment of scleroderma.

Background:

There are two subtypes of systemic scleroderma: diffuse and limited (2). Limited skin involvement includes skin involvement distal to the elbows and knees and may include the neck and face, but spares the trunk and proximal extremities. Diffuse scleroderma has more extensive skin involvement including trunk or proximal extremities and is associated with more internal organ involvement and increased mortality (4). For instance, significant interstitial lung disease, cardiomyopathy and scleroderma renal crisis are more common in diffuse scleroderma than limited. The extent of organ involvement in these areas may correlate with the extent of skin involvement and worsening skin involvement is associated with increased mortality and worse overall health function as measured by the Health Assessment Questionnaire (HAQ) (5).

Formulation of Objective:

Various signals that could be therapeutically down regulated in scleroderma such as PDGF, VEGF, endothelin, and TGFβ are potential therapeutic targets. The inhibition of tyrosine kinase can decrease cell growth and could be a key signal modifier in scleroderma (6). Signal transduction modification with selected targets has been very successful in the treatment of some cancers, such as using Gleevec in chronic myelocytic leukemia (7).

Gleevec (imatinib) is an oral tyrosine kinase inhibitor. It is used in the treatment of CML and some GI stromal tumors, with a reduction in mortality in CML. Tyrosine kinase activates PDGF and TGFbeta, which are key signals in scleroderma so a proof of concept study is needed to determine if there is a biological signal to proceed in a disease of fibrosis such as scleroderma. PDGF regulation is important in fibrotic diseases by stimulating replication and migration of myofibroblasts (8).

Protocol:

Subjects with active diffuse scleroderma will be enrolled after consenting and will receive Gleevec 400mg/od or placebo. Serum and skin biopsies will be collected for biomarkers. Serum samples will be taken at baseline, 3 and 6 months and analyzed by ELISA/multiplexing for changes in profibrotic cytokines including PDGF, VEGF, endothelin, and TGFβ. Skin biopsies will be taken prior to the first dose and at 6 months. Modified Rodnan Skin Score (MRSS), Health Assessment Questionnaire (HAQ), MD and patient global assessments will also be done at times 0, 3, and 6 months. SF36 and Health Transition Score will be done at 0 and 6 months. Biochemistry for safety and inflammation will be done once a month for the duration of the trial.

Gleevec at 400 mg/od or placebo will be given orally with food and a large glass of water for 6 months. As this is a proof of concept and Phase IIa trial they will be randomized into active vs. placebo groups in a 4:1 ratio, where n=20. Therefore, 16 patients will receive active drug and 4 will receive placebo.

Specific Aims:

1. Primary outcome measurement: changes in cytokine expression in skin biopsies and serum samples for profibrotic cytokines.
2. To determine the between groups differences from baseline to final skin score on Gleevec and placebo at 6 months using the Modified Rodnan Skin Score (MRSS).
3. To compare the AEs (adverse events) and SAEs (serious adverse events) between the groups.
4. Secondary objectives will be:

Comparing secondary outcome measurements such as: MD global, patient global, HAQ, SF36, Health Transition, ESR, CRP.

Randomization and Blinding:

The randomization will be stratified by current use of methotrexate. It is anticipated that the majority of patients in this trial will not be taking methotrexate at time of randomization, but stratification should balance the groups if there is a heterogenous response. The randomization will be done in balanced blocks of 5, after stratification by methotrexate use. The pharmacy will be called and will provide the medication and will have the randomization code. The trial is blinded where the patient, the research nurse performing study procedures including dispensing the study drug, and the physician doing the outcome assessments will all be unaware of treatment allocation.

Concomitant Medications:

Stable dose concomitant methotrexate of up to 25 mg/week if tolerated (po or sc) can be continued throughout the study. In addition, if necessary, folate can be added or increased to decrease side effects.

All standard of care is allowed except for the medications listed above. Thus treatment for GERD, Raynaud's, digital ulcers, HTN, delayed GI emptying, small bowel overgrowth, Sjogren's symptoms, arthritis (using NSAIDs or low dose prednisone) is allowed. Severe PAH and severe ILD is excluded as there could be expectations that this comorbidity may interfere with the current 24-week treatment protocol. Steroids can be increased in the rare chance that a patient develops a complication or co-morbidity that requires higher doses of steroids as part of standard care. Regular need for antibiotics for small bowel overgrowth is allowed.

Good clinical practice will be followed and other appropriate treatment will not be denied. This is an 'add-on' treatment to standard care. Concomitant medications will be assumed to be held stable throughout the study. Patients taking any medications that may interact with Gleevec (eg. SSRIs, TCA, trazadone, benzodiazepines, betablockers, etc.) will be monitored cautiously.

Since Gleevec has been postulated (by a case report) to improve pulmonary arterial hypertension (PAH) annual echocardiograms that are done as part of standard care may be compared between the groups determining the estimated PAP on echocardiogram (9).

AEs and SAEs:

The University of Western Ontario Ethics Committee will approve the protocol and any amendments and will be informed of any SAEs as per usual research conduct. The patients are free to withdraw consent or drop out at any time with no adverse effect on their future care. As per any trial, AEs and SAEs will be collected. SAEs will be reported in an expedited way to the UWO Ethics Committee and Novartis.

Pregnancies:

Pregnancy or fathering of a child, although not itself a serious adverse event, should also be reported on a serious adverse event form or pregnancy form and be followed up to determine outcome, including spontaneous or voluntary termination, details of birth, and the presence or absence of any birth defects or congenital abnormalities. In addition to any pregnancy or fathering of a child within 84 days (12 weeks or 3 months) after the last Gleevec intake has to be reported and recorded as an SAE.

Any pregnancy that occurs during study participation should be reported using a Clinical Trial Pregnancy Form. To ensure patient safety each pregnancy must also be reported to Novartis within 24 hours of learning of its occurrence. The pregnancy should be followed up to determine outcome, including spontaneous or voluntary termination, details of birth, and the presence or absence of any birth defects or congenital abnormalities or maternal and newborn complications.

Patients will be informed of the risks involved in becoming pregnant while taking Gleevec in the Letter of Information and female partners of male study participants will be required to read and sign a "Pregnant Partner Data Release Form" acknowledging that they have been informed of these risks as well.

Discontinuation of Treatment:

The patients are free to drop out at any time. A severe allergic reaction will necessitate withdrawal. If there are sustained cytopenias (WBC <2.0, Hbg < 8.0 or Plt < 50,000) for 2 infusions in a row then the patient will be withdrawn. If there is a WBC < 1.0 or Hbg < 7.5 or Plt < 10,000 at any time, the patient will be withdrawn. If there are sustained elevations of AST/ALT twice in a row, of twice the upper limit of normal, then the methotrexate will be decreased by 5 mg/week. If the elevation persists for 2 more tests, the methotrexate will be held for two weeks and the liver enzymes repeated. If still elevated, the methotrexate will be cut in half and if still elevated and no other concomitant meds are thought to be causing the elevation, then the patient will be withdrawn.

Sample Size:

This study is a pilot and is not anticipated to have enough power to have a statistically significant between groups difference on skin score. However, the effects on fibrosis and other mediators in serum and tissue specimens may help to determine if a larger trial should be a 'go' or 'no go'.

Analysis:

This will be a modified intent to treat analysis, where any patient receiving at least one dose of the study drug will be analyzed, and for dropouts the last observation will be carried forward (LOCF). The primary outcome measurement will be changes in profibrotic cytokine expression in serum and urine samples and skin biopsies. Multiplexing will be used to measure up to 30 analytes of interest in one 50ul sample of any biological fluid. Statistics will include the between groups (active and placebo) difference at 24 weeks (6 months) in the MRSS. There will be a between groups assessment of HAQ, ESR and CRP for placebo compared to Gleevec. The SF36 and Health Transition Scores will be compared using paired tests. AEs and SAEs will be quantified and compared between placebo and active treatment. PK and PD data will only be analyzed if there is a thought of continuing drug development in this area. If the data appear to demonstrate some benefit, then a repeated measures ANOVA will be done to determine if there are between groups differences at various time points.

Data Safety Monitoring Board:

All SAEs will be reported to the Ethics Committee and to Novartis. An independent safety board blinded to treatment allocation will meet at 3 months to monitor study progress and SAEs. There will be no interim analysis, as the study is not powered to do one. Safety events will be collected up until one month after discontinuing study drug in all cases wherever possible.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to give informed consent.
* Subjects must meet preliminary criteria for scleroderma.
* Subjects must have diffuse skin involvement.
* Disease must appear to be active as measured by worsening skin score and/or increased ESR.
* Serum SGOT < 1.5 times upper limit of normal.
* Bilirubin < 1.5 times upper limit of normal.
* AST/ALT < 2.5 times upper limit of normal

Exclusion Criteria:

* Any past exposure to Gleevec.
* Women of child bearing potential must be practicing an acceptable form of contraception (OCP, depo-provera, IUD, condoms with spermicidal or sterilization of subject or partner).
* Women who are breastfeeding.
* Men whose partners could conceive must be practicing acceptable contraception (see above).
* Certain abnormal labs including: Neutrophil count <1.5X109/L, platelets < 50X109/L.
* Serious comorbidity that may impair the ability to complete the study (such as severe heart disease, severe pulmonary hypertension) and other comorbidities.
* Prednisone at doses of >10mg/od.
* Other potential disease modifying drugs such as cyclophosphamide, mycophenylate and methotrexate.
* Serious liver disease.
* Creatinine >200.
* Excluded: Ketoconazole and fluconazole, cyclosporine, rifampin, phenytoin nefazodone, pimozide, propafenone, quinidine, sibutramine and sildenafil where drug interactions could occur.
* Subjects taking endothelin receptor blockers such as bosentan and sitaxsentan.
* Alcohol consumption of > 3 drinks per week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Changes in the levels of fibrotic and inflammatory biomarkers in plasma samples. | Plasma samples were taken at baseline (0), 3 and 6 months (study end).
  Twenty-six fibrotic and inflammatory biomarkers were measured: PDGF-AA, PDGF-AB/BB, IL-13, IL-17, VEGF, TGF-beta1, sVCAM-1, sICAM-1, sE-selectin, MMP-9, tPAI-1, IL-1alpha, IL-1 beta, IL-4, IL-6, IL-10, IL-12p70, IL-13, TNF- alpha, sCD40L, IFN- gamma, MCP-1, MCP-3, MIP-1 alpha, MIP-1 beta, and chemokine ligand 5 (CCL5 - also known as RANTES). Biomarkers were measured using multiplexed immunoassays (Millipore Corp., MA) and ELISA for TGF- beta 1 (BD Biosciences, NJ).
Changes in the levels of fibrotic and inflammatory biomarkers in skin biopsies. | Baseline and 6 months (study end).
  Twenty-six fibrotic and inflammatory biomarkers were measured: PDGF-AA, PDGF-AB/BB, IL-13, IL-17, VEGF, TGF-beta1, sVCAM-1, sICAM-1, sE-selectin, MMP-9, tPAI-1, IL-1alpha, IL-1 beta, IL-4, IL-6, IL-10, IL-12p70, IL-13, TNF- alpha, sCD40L, IFN- gamma, MCP-1, MCP-3, MIP-1 alpha, MIP-1 beta, and chemokine ligand 5 (CCL5 - also known as RANTES). Biomarkers were measured using multiplexed immunoassays (Millipore Corp., MA) and ELISA for TGF- beta 1 (BD Biosciences, NJ).

SECONDARY OUTCOMES:
Modified Rodnan Skin Score (MRSS) | Baseline, 3 months and 6 months (study end).
  The Modified Rodnan Skin Score (MRSS) is a validated outcome measurement and is the usual primary outcome measurement for all trials of disease modification in scleroderma. It is positively correlated with internal organ involvement and has been shown to improve or worsen in many patients.
Adverse events and serious adverse events | From treatment start until 4 weeks after after the patient has stopped study participation
  This study will use the CTCAE (NCI Common Terminology Criteria for Adverse Events) versions 3.0 for toxicity and adverse event reporting. If multiple dose-reducing toxicities are present, the greatest dose reduction schedule should be used. Information about all adverse events will be collected and recorded on the Adverse Event Case Report Form and followed as appropriate. Serious adverse events occurring more than 4 weeks after study discontinuation need only be reported if a relationship to the study drug (or therapy) is suspected.
Health Assessment Questionnaire | Baseline, 3 months and 6 months (study end).
Patient Global Assessment | Baseline, 3 months and 6 months (study end).
  Patient assessment of global disease activity on a 100 mm visual analog scale.
Physician Global Assessment | Baseline, 3 months and 6 months (study end).
  Physician global assessment of disease activity on a 100 mm visual analog scale.
The Short Form (36) Health Survey | Baseline and 6 months.
Health Transitiion Score | Baseline and 6 months.
  "Compared to 6 months ago, how do you rate your health overall?: Much worse, worse, same, better, much better".

CONTACTS AND LOCATIONS:
Overall Officials: Janet E Pope, MD MPH FRCPC, Principal Investigator — Lawson Health Research Institute, Western University
Locations (1):
- Lawson Health Research Institute, London, Ontario, Canada

REFERENCES:
- [Background] Nadashkevich O, Davis P, Fritzler MJ. A proposal of criteria for the classification of systemic sclerosis. Med Sci Monit. 2004 Nov;10(11):CR615-21. Epub 2004 Oct 26. PMID 15507853
- [Background] LeRoy EC, Black C, Fleischmajer R, Jablonska S, Krieg T, Medsger TA Jr, Rowell N, Wollheim F. Scleroderma (systemic sclerosis): classification, subsets and pathogenesis. J Rheumatol. 1988 Feb;15(2):202-5. No abstract available. PMID 3361530
- [Background] Thompson AE, Pope JE. Increased prevalence of scleroderma in southwestern Ontario: a cluster analysis. J Rheumatol. 2002 Sep;29(9):1867-73. PMID 12233880
- [Background] Haugeberg G, Brodin C, Johnsen V. [Systemic sclerosis. A rare connective tissue disease with manifestations in many organs]. Tidsskr Nor Laegeforen. 1995 Nov 30;115(29):3619-21. Norwegian. PMID 8539716
- [Background] Fries JF, Spitz P, Kraines RG, Holman HR. Measurement of patient outcome in arthritis. Arthritis Rheum. 1980 Feb;23(2):137-45. doi: 10.1002/art.1780230202. PMID 7362664
- [Background] Lankat-Buttgereit B, Horsch D, Barth P, Arnold R, Blocker S, Goke R. Effects of the tyrosine kinase inhibitor imatinib on neuroendocrine tumor cell growth. Digestion. 2005;71(3):131-40. doi: 10.1159/000084647. Epub 2005 Mar 22. PMID 15785039
- [Background] Newell DR. How to develop a successful cancer drug--molecules to medicines or targets to treatments? Eur J Cancer. 2005 Mar;41(5):676-82. doi: 10.1016/j.ejca.2004.12.024. PMID 15763642
- [Background] Bonner JC. Regulation of PDGF and its receptors in fibrotic diseases. Cytokine Growth Factor Rev. 2004 Aug;15(4):255-73. doi: 10.1016/j.cytogfr.2004.03.006. PMID 15207816
- [Background] Ghofrani HA, Seeger W, Grimminger F. Imatinib for the treatment of pulmonary arterial hypertension. N Engl J Med. 2005 Sep 29;353(13):1412-3. doi: 10.1056/NEJMc051946. No abstract available. PMID 16192491
- [Derived] Pope J, Walker KM, de Leon F, Vanderhoek L, Seney S, Summers KL. Correlations between changes in cytokines and clinical outcomes for early phase (proof of concept) trials in active diffuse systemic sclerosis using data from an imatinib study. Rheumatology (Oxford). 2014 Oct;53(10):1830-4. doi: 10.1093/rheumatology/keu216. Epub 2014 May 20. PMID 24850877